CLINICAL TRIAL: NCT04853979
Title: Awake Prone Positioning in COVID-19 Suspects With Hypoxemic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Tim Richard Edmund Harris, Vice chairman Education Emergency Department, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-01-20-1227
Record Dates: First submitted 2021-04-12; First posted 2021-04-22 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Patients; Hypoxemic Respiratory Failure; Prone Position
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Masking Description: Prone position cannot be masked to any member in the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRONE (Experimental): Any combination of prone or side position for 3 hours, 3 times a day for 3 days.
  Interventions: Other: PRONE POSITION
- NO PRONE (Active Comparator): Usual care
  Interventions: Other: PRONE POSITION

INTERVENTIONS:
Other: PRONE POSITION — Any combination of prone or side position for 3 hours, 3 times a day for 3 days

SUMMARY:
The investigator hypothesis is that early implementation of early, awake prone position for patients with COVID-19 pneumonia requiring oxygen therapy will reduce the need for escalation of respiratory support. Escalation of respiratory support is defined as the need for respiratory support with HFNO, NIV or IV.

DETAILED DESCRIPTION:
The world health organization has designated the Severe Acute Respiratory Syndrome coronavirus 2 (SARS-CoV-2) as an ongoing pandemic and a public health emergency of international concern. The disease is estimated to be severe in 20% of patients and about 5-10% will need critical care with respiratory support. ARDS is thought to be the main cause of respiratory failure in COVID-19 patients. Research is still ongoing to further elucidate the different ARDS subtypes that may exist in COVID-19. It is crucial to find new targets for treatment and support of COVID-19 patients with respiratory failure.

Prone positioning causes a substantial improvement in oxygenation that appear to persist after the patient is returned to a supine position. It has also been shown to have a significant mortality benefit in invasively ventilated ARDS patients. Observational studies have shown improvement in oxygenation with awake prone positioning in non-intubated patients with COVID-19 pneumonia. There is no published RCTs to date. It remains unclear whether prone positioning averts invasive or non-invasive ventilation, accelerates recovery, or reduces mortality. Similarly, there is no data on presumed viral pneumonia. Future studies are needed to identify the optimal indications for, duration of pronation, and assessment of response.

Hypothesis: The investigator hypothesis is that early implementation of early, awake pronation for patients with Covid19 pneumonia requiring oxygen therapy will reduce the need for escalation of respiratory support. Escalation of respiratory support is defined as the need for respiratory support with HFNO, NIV or IV Research participants: Adults 18 years and older with suspected or confirmed COVID-19 presenting to HMC with hypoxemic respiratory failure (PF<200 or SpO2 less than 94% on FiO2>=0.4 or =>5 lit/min O2)

Design: This is a non-blinded randomized controlled trial. Participants will be randomized to one of two study arms:

1. Intervention arm: Any combination of prone or side position (defined as any part of the anterior chest wall being in contact with the bed) for at least 3 hours and up to 16 hours per day during wakefulness. Patients will be asked to prone on three occasions: morning, afternoon and evening. Breaks of 30-120 min are allowed in sitting position or supine each 4 hours. Bed elevation of >30 degrees will be maintained unless otherwise requested by the patient. No control or intervention is made during sleep periods. Intervention will last for up to 3 days or until the patient achieves oxygen saturations of 94-98% on room air. Oxygen delivery may be via NC, HM, HFNC or NIV.
2. Control arm: Usual care (no Prone unless asleep and assumes this position spontaneously). The patient is able to adopt their preferred natural position. The bed will be elevated >30 degrees unless requested otherwise by the patient. However prone position may be used as rescue therapy if oxygen requirements are =>15 lit/min O2 or HFNC/NIV with FiO2 =>0.6 with O2 saturation less than 90% at the discretion of the treating physician.

Methods and outcomes:

Data will be analyzed for escalation of respiratory support within the first three days of the study. Escalation of respiratory support is defined as follows:

* escalation from NP/HC/NRB to HFNO or NIV or IV
* escalation from HFNO or NIV to IV Several secondary outcomes will be analyzed as well as outlined in outcomes section.

Based on previous studies of prone position in COVID-19 patients, anticipate an improvement in oxygenation and possible prevention of intubation with shorter mechanical ventilation times. Awake proning has been shown to be safe in local practice.

ELIGIBILITY:
Inclusion Criteria: - All adults with suspected or confirmed COVID-19 and hypoxemia respiratory failure.

* SPO2 less than 94% or Oxygen requirment of more than 5 liters.
* Requiring oxygen therapy in Hospital< 24 hours

Exclusion Criteria:

* Clinical assessment for immediate intervention.
* PF<50
* SF<90
* RR>60bpm
* Hemodynamics instability with need for vasopressors.
* MSOF
* Age<18
* Pregnancy
* Impaired LOC, agitation or lack of cooperative patient.
* BMI>40
* Unstable spine or pelvis
* Abdominal wound
* Pnemothorax
* Any injury or illness that may be worsened or result in pain as a result of prone position.
* DNAR
* Any contraindicaton to prone position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients requiring escalation to NIV (CPAP or BIPAP) or IV in each group | 30 days
  To assess the potential for prone position to reduce the requirement for escalation of respiratory support.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harris TRE, Bhutta ZA, Qureshi I, Kharma N, Raza T, Hssain AA, Pathare AS, D'Silva A, Khatib MY, Mohamedali MGH, Macineira IMG, Garcia Hernandez VR, Garcia JR, Thomas SH, Pathan SA. A randomised clinical trial of awake prone positioning in COVID-19 suspects with acute hypoxemic respiratory failure. Contemp Clin Trials Commun. 2024 Apr 13;39:101295. doi: 10.1016/j.conctc.2024.101295. eCollection 2024 Jun. PMID 38689829